CLINICAL TRIAL: NCT06588244
Title: Ischemia in Patients with Non- Obstructive Disease (INOCA) - a Local Prospective Registry (INOCA-Naples)
Brief Title: INOCA-NA a Local Prospective Registry
Acronym: INOCA-NA
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luigi Di Serafino, Principal Investigator, Clinical Professor, Federico II University
Other Study IDs: 160/2024
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Ischemia, Myocardial; Non-Obstructive Coronary Atherosclerosis; Microcirculatory Status; Coronary Microvascular Dysfunction (CMD)
Keywords: INOCA; CMD; VSA
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- INOCA: Patients presenting with symptoms or signs of myocardial ischemia with non-obstructing coronary artery disease

SUMMARY:
The present study has the following objectives:

1. To investigate the prevalence of INOCA in patients referring for a clinically indicated coronary angiography (CA) c/o Division of Cardiology - Federico II University Hospital;
2. To stratify in INOCA endotypes patients according to the presence or absence of alternative (i.e. non obstructive CAD) causes of myocardial ischemia detected during CA clinically indicated through physiology tests;
3. to implement a stratified therapy in these patients considering the different INOCA endotypes and evaluate the impact on angina class and quality of life as well as cardiac hospitalization and coronary revascularization during 5 year follow up

DETAILED DESCRIPTION:
Eligible patients with angina and/or positive stress test undergoing clinical indicated CA detecting non-obstructive CAD will be studied as follows:

* Functional evaluation by fractional flow reserve (FFR), instantaneous wave-free ratio (iFR), Resting Full-Cycle Ratio (RFR) of any stenosis that is angio- graphically considered > 50%;
* In case of stenosis <50% or >50% but with negative functional evaluation (FFR >0.80 and iFR/RFR

  >0.90), coronary flow reserve (CFR) and index of microvascular resistance (IMR) will be performed. IMR and CFR will be evaluated, using an intracoro- nary wire;
* In case of CFR>2.0 and IMR<25, acetylcholine test will be performed. Intracoronary acetylcholine (ACh) will be administrated to detect epicardial (fo- cal or diffuse) or microvascular spasm.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation of chronic ischemic heart dis- ease (IHD), requiring coronary angiography for the diagnosis;
* Absence of obstructive coronary artery disease (CAD) at coronary angiography;
* Age > 18 years.
* Ability to provide a valid informed consent to the study procedure at the time of baseline evaluation;

Exclusion Criteria:

Clinical presentation of acute coronary syndrome (ACS) or cardiogenic shock;

* Presence of obstructive CAD with at least 1 significant coronary artery stenosis, defined as diameterstenosis >50% and FFR ≤0.80 (or iFR/RFR ≤0.89);
* Previous coronary artery bypass grafting (CABG);
* Left ventricular systolic dysfunction, defined as ejection fraction (EF) <40%;
* Severe valvular heart disease;
* Pregnant or breastfeeding women
* Known hypersensitivity or contraindication to any of the drugs used for coronary physiology testing (adenosine, nitrates, acetylcholine)
* Inability or unwillingness to provide a valid in- formed consent to the study procedure at the time of baseline evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting with signs or symptoms potentially related to myocardial ischemia and requiring a functional coronary angiography for specific diagnosis will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
MACE | 12 and 60 months
  Occurrence of Cardiovascular death, Myocardial infarction, Coronary revascularization
Degree of Angina | 12 and 60 months
  The degree of angina will be assessed using The Seattle Angina Questionnaire - 7 (SAQ-7) contains 7 questions used to measure health status in patients with coronary artery disease (CAD). The score is generated for each domain and it is scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status.
QoL | 12 and 60 months
  Quality of life will be assessed using the 5-level EuroQoL 5-dimensions Questionnaire (EQ-5D-5L). The EQ-5D-5L descriptive system comprises the same five dimensions as the EQ-5D-3L (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN/DISCOMFORT and ANXIETY / DEPRESSION), but each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each of the five dimensions. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. An EQ-5D health state is deemed to be 'better' than another if it is better on at least one dimension and is no worse in any other dimension. An EQ-5D health state is deemed to be 'worse' than another if it is worse in at least one dimension and is no better in any other dimension.

OTHER OUTCOMES:
TIMI Frame Count | up to 24 hours
  To evaluate the accuracy of TIMI Frame Count (TFC) to identify specific INOCA endotypes. TFC will be evaluated dunring invasive assessement before and after administration of nitrates. Patients with different INOCA endotypes will be compared in terms of TFC.
EndoPAT_Endoscore | 1 day and 12 months
  To evaluate whether the assessment of peripheral microcirculation, as assessed with EndoPAT test might be useful to identify specific INOCA endotypes. The EndoPAT detects plethysmographic pressure changes in the finger tips caused by the arterial pulse and translates this to a peripheral arterial tone (PAT). We will evaluate the Endoscore which has been previosly reported to be significantly decreased in patients with coronary artery disease, thereby the lower the endoscore the higher the risk of endothelial dysfunction.
EndoPAT_RH | 1 day and 12 months
  To evaluate whether the assessment of peripheral microcirculation, as assessed with EndoPAT test might be useful to identify specific INOCA endotypes. The EndoPAT detects plethysmographic pressure changes in the finger tips caused by the arterial pulse and translates this to a peripheral arterial tone (PAT). We will evaluate the Reactive Hyperemic Index (RHI) which has been found to be significantly decreased in patients with coronary artery disease, thereby the lower the RHI values the higher the risk of endothelial dysfunction.
Nitrates effects on CFR | up to 5 minutes
  To evaluate any changes in terms of hemodynamic parameters after i.c. administration of nitrates, which is normally administered during the invasive functional coronary angiography. In particular, we will evaluate the Coronary Flow Reserve (CFR), measured as the ratio between the mean transit time at rest and the mean transit time during maximal hyperemia.
Nitrates effects on MMR | up to 5 minutes
  To evaluate any changes in terms of hemodynamic parameters after i.c. administration of nitrates, which is normally administered during the invasive functional coronary angiography. In particular, we will evaluate the Microvascular resistance reserve (MRR), measured as the ratio between the CFR and the fractional flow reserve (FFR) corrected for driving pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- DPT of Advanced Biomedical Sciences, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Privacy concerns